CLINICAL TRIAL: NCT04607265
Title: Channel Detection to Predict Ventricular Arrhythmia in Patients With Non-ischemic Cardiomyopathy
Brief Title: Sudden Death Stratification
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0838
Record Dates: First submitted 2020-09-28; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-09

CONDITIONS: Non-ischemic Cardiomyopathy
Keywords: LGE MRI; Ventricular tachycardia; sudden cardiac death; non-ischemic cardiomyopathy
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ventricular tachycardia (VT) group: NICM patients admitted for a VT ablation with a pre-operative cardiac- MRI.
  Interventions: Diagnostic Test: Cardiac MRI
- Control group: NICM patients without ventricular arrhythmia and a previous cardiac-MRI. The matching with the VT group was based on the age of the patients, the mean LVEF, the time between the initial diagnosis and the MRI examination, and the origin of the NICM.
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Comparison of scar characteristics on cardiac MRI between the two groups.

SUMMARY:
Sudden cardiac death (SCD) risk stratification is a challenge in non-ischemic cardiomyopathy (NICM). The underlying mechanism of monomorphic ventricular tachycardia (VT) is mostly scar related. While electrophysiological mechanisms underlying ventricular arrhythmia are well known, late gadolinium enhanced (LGE) cardiac MRI-3D reconstructions are now able to guide VT ablation procedures. Such exam may help in identifying specific properties of scar at risk of malignant arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Adult with NICM
* Previous history of ventricular tachycardia (VT) and no previous history of VT

Exclusion Criteria:

* Inherited cardiomyopathies
* Previous history of myocarditis WITHOUT oedema/scar at the MRI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that underwent VT ablation, had a cardiac MRI prior to the ablation and suffered from non-ischemic cardiomyopathy (NICM) were included in the VT group. A 2:1 ratio of patients with non-ischemic cardiomyopathy and no history of ventricular tachycardia were included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Detect pro arrhythmogenic scar characteristics | baseline : collected at the time of the cardiac MRI
  The outcomes will aim to provide scar characteristics from 3D cardiac MRI reconstructions to detect pro arrhythmic properties in NICM patients. Comparisons between NICM patients who experienced VT ablation and NICM patients without history of ventricular arrhythmia will be made.
  In both groups, Primary outcome will aim to measure the number of the conducting channels into scars (n).